CLINICAL TRIAL: NCT01429220
Title: Automated Parkinson's Disease (PD) Motor Symptom Assessment for Deep Brain Stimulation (DBS) Programming
Status: Completed | Type: Observational
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 5R44AG033520-03 (NIH)
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson's Disease
Keywords: deep brain stimulation; monopolar review; motion sensors; tremor; bradykinesia
MeSH Terms: conditions — Parkinson Disease; Tremor; Hypokinesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the utility of a portable motion sensor-based system designed to assist with deep brain stimulation (DBS) programming sessions for Parkinson's disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr stage 2 or worse when off medications
* Average tremor and/or bradykinesia Unified Disease Rating Scale (UPDRS) score greater than 2 off meds
* L-dopa responsive with clearly defined "on" periods, UPDRS motor III average tremor and bradykinesia improves by 25%
* Stable on medical therapy for at least one month prior to study enrollment
* Clinical approval to undergo unilateral DBS surgery targeting the STN or GPi
* Available to participate for six months following DBS surgery

Exclusion Criteria:

* "Parkinson's plus" syndromes, secondary, or atypical Parkinson's syndromes (e.g. progressive supranuclear palsy, striato-nigral degeneration, multiple system atrophy, post-stroke, post-traumatic, or post-encephalitic Parkinson's. These patients have cardinal symptoms characteristic of PD but with additional symptoms indicating other organic brain dysfunction, such as gaze palsies, autonomic dysfunction, lack of response to L-dopa, these individuals tend not to improve with standard treatments for PD)
* previous Parkinson's Disease surgery
* medical contraindications to surgery or stimulation (e.g. uncontrolled hypertension, advanced coronary artery disease, other implanted stimulation or electronically-controlled devices including cardiac demand pacemaker, aneurysm clips, cochlear implants, or a spinal cord stimulator) (Note: for the subject who receives either a pacemaker and/or defibrillator after this study enrollment, he/she will be allowed to continue the study if the neurostimulator system can be adequately programmed to permit system compatibility)
* contraindication to magnetic resonance imaging (e.g. indwelling metal fragments or implants that might be affected by MRI)
* neuropsychological dysfunction (e.g. dementia) that would contraindicate surgery
* intracranial abnormalities that would contraindicate surgery (e.g. stroke, tumor, vascular abnormality affecting the target area)

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-08; Primary Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States